CLINICAL TRIAL: NCT03671005
Title: Mindfulness-based Group Therapy for Inpatients With Schizophrenia Spectrum Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to covid restrictions the recruitment for this study has been paused after the feasibility and acceptability data was published.
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kerem Böge, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APS2018
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Psychotic Disorder
MeSH Terms: conditions — Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A single-centered randomized controlled trial with a parallel-groups design is utilized, comprising of mindfulness-based group therapy (MBGT) in addition to treatment as usual (TAU) in the experimental condition, and TAU in the control condition
Who Masked: Outcomes Assessor
Masking Description: A blinded psychiatrist who works independently of the (co-) therapist conducts the rater-questionnaires. Due to the psychotherapeutic nature of the study, information about the treatment allocation has to be shared with the co-therapist and the participants. Randomization is conducted by the Random Group Generator (pubmed, 2018).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based group therapy (MBGT) (Experimental): The mindfulness-based group therapy (MBGT) involves a four-week manual with three group therapy sessions per week in addition to TAU. The therapy represents the first German group-based mindfulness manual for psychosis. One sixty-minute session was held by a certified psychotherapist who is experienced in mindfulness-based therapy. A trained co-therapist implements two 30-minute sessions. On a weekly basis, a new theme is discussed in the three sessions to ensure the internalization of different mindfulness concepts. Namely, the topics Mindfulness of the Breath (1), Mindfulness of the Senses in the Context of Nature (2), Mindfulness of Detachment (3), and Mindfulness in the Context of Bodily Awareness (4) are addressed during the group-sessions.
  Interventions: Behavioral: Mindfulness-based group therapy
- treatment as usual (TAU) (Active Comparator): Treatment as usual (TAU) at the ward consists of a variety of daily activity groups the patients can choose from. Every patient at the ward receives a daily schedule depending on individual needs for therapy. The therapies offered at the ward include occupational therapy, physiotherapy, psychoeducative groups, and concentration practice of two levels, all not related to mindfulness interventions. In addition to the group activities at the ward, every patient receives individual psychotherapy sessions at least once a week, held by a certified psychiatrist or psychologist. Psychopharmacological treatment is provided by the physicians, and social workers are available in order to support patients in managing their everyday lives after the stationary treatment. Weekly group meetings at the ward, together with the treating physicians, psychotherapists, social workers and the respective patient, foster the exchange success and possible improvements of the treatment.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Mindfulness-based group therapy — see above
  Arms: Mindfulness-based group therapy (MBGT)
Other: Treatment as usual — see above
  Arms: treatment as usual (TAU)

SUMMARY:
A single-centered randomized controlled trial with a parallel-groups design is utilized, comprised of mindfulness-based group therapy (MBGT) in the experimental condition, and treatment as usual (TAU) in the control condition. Participants in the experimental condition continued their regular psychiatric treatment (TAU) next to the participation in the MBGT. In order to evaluate possible psychotherapeutic effects, self-report and other clinical questionnaires including interviews and app-based assessments are evaluated before (T0), and after the four-week intervention (T1).

Ward psychiatrists identify eligible participants and invite them to participate in the study. An eligibility screening is held by the study assistant at baseline, introducing the study, providing informed consent in written form, as well as conducting the self-report measures and app-based assessments. A blinded psychiatrist who works independently of the (co-) therapist conducts the remaining rater-questionnaires. Due to the psychotherapeutic nature of the study, information about the treatment allocation had to be shared with the co-therapist and the participants. Randomization was conducted by the Random Group Generator (pubmed, 2018). The data management plan includes standard procedures for data-handling such as using anonymized identification codes for patient data. The participants have the right to access their data, and the right to claim an annihilation. The data is being stored in locked cupboards, only allowing researchers involved in the study to access the data.

ELIGIBILITY:
Inclusion criteria:

* male and female participants
* treated as psychiatric inpatients at the psychosis - or social-psychiatric day ward
* between 18 and 65 years of age
* diagnosis of a schizophrenia-spectrum disorder according to the Diagnostical and Statistical Manual 5th edition) and the International Statistical Classification of Diseases and Related Health Problems(ICD-10) code F2
* ability to give informed consent
* willingness and ability to engage in psychotherapeutic group therapy
* low to moderate psychotic state indicated with a score of 6 < for each item at the Positive scale of the Positive and Negative Syndrome Scale (PANSS, Peralta & Cuesta, 1994)

Exclusion criteria:

* a score ≥ 6, suggesting an acute psychotic episode with severe psychotic symptoms (Peralta& Cuesta, 1994)
* acute suicidality, assessed by item eight of the Calgary Depression Scale for Schizophrenia > 1 (Addington, Addington, Maticka-Tyndale, & Joyce, 1992)
* any neurological disorders that may affect cognitive functioning
* acute substance abuse other than nicotine and prescribed medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
mindfulness | 6 months
  The Freiburg Mindfulness Inventory (FMI) to measure mindfulness, 14 items on a scale from 1 - 4 (1 = seldom, 4 = almost always)
mindfulness | 6 months
  Comprehensive Inventory of mindfulness experience (CHIME, 37 items on a scale from 1 (almost never) to 6 (almost always)
mindfulness | 6 months
  Southampton mindfulness questionnaire (SMQ), 16 items on a scale from 1 (applies fully) to 7 (does not apply at all)

SECONDARY OUTCOMES:
broad cognitive functioning | 6 months
  CANTAB mobile App to assess cognitive functioning, validated version for schizophrenia
personal and social performance | 4 weeks
  Personal and Social Performance Scale (PSP), Interview measures personal and social functioning in the domains of: Socially useful activities (eg, work and study), Personal and social relationships, Self-care, Disturbing and aggressive behaviors. Different domains are rated on a scale from absent to highly severe.
Symptom - Depression | 6 months
  Calgary Depression-Scale for Schizophrenia measures depressive symptoms based on 9 items rated on a scale from absent to severe.
symptomatology - positive and negative symptoms | 4 weeks
  Positive and Negative Syndrome Scale (PANSS) to assess symptoms on a scale from 1 (non-existent) to 7 (extremely severe, 14 questions
Symptoms - Depression and Anxiety | 6 months
  Depression Anxiety Stress Scales (DASS), 21 questions that can be answered on a scale from 0 (does not apply to me) to 3 (applies to me strongly/most of the time)
cognitive fusion | 6 months
  Cognitive Fusion Questionnaire (CFQ), 7 questions that can be answered on a scale from 1(not applicable) to 7 (applies always)
psychological flexibility | 6 months
  Acceptance and Action Questionnaire (AAQ-II) measures psychological flexibility. 7 questions that can be measured on a scale from 1 (never true) to 7 (always true)
Quality of Life - domains assessed include physical and psychological health, social relationships and environment | 6 months
  World Health Organisation Quality of Life (WHO-QOL-Bref) to assess quality of life measured on a scale from 1 (never) to 5 (always). Facets incorporated in the 4 domains: 1. Physical health - Activities of daily living Dependence on medicinal substances and medical aids Energy and fatigue Mobility Pain and discomfort Sleep and rest Work Capacity; 2. Psychological - Bodily image and appearance Negative feelings Positive feelings Self-esteem Spirituality / Religion / Personal beliefs Thinking, learning, memory and concentration; 3. Social relationships - Personal relationships Social support Sexual activity; 4. Environment - Financial resources Freedom, physical safety and security Health and social care: accessibility and quality Home environment Opportunities for acquiring new information and skills Participation in and opportunities for recreation / leisure activities Physical environment (pollution / noise / traffic / climate) Transport.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boge K, Hahne I, Bergmann N, Wingenfeld K, Zierhut M, Thomas N, Ta TMT, Bajbouj M, Hahn E. Mindfulness-based group therapy for in-patients with schizophrenia spectrum disorders - Feasibility, acceptability, and preliminary outcomes of a rater-blinded randomized controlled trial. Schizophr Res. 2021 Feb;228:134-144. doi: 10.1016/j.schres.2020.12.008. Epub 2021 Jan 9. PMID 33434727
- See also: app-based assessment — http://www.cambridgecognition.com/cantab/